CLINICAL TRIAL: NCT02084173
Title: Motivational Enhancement Therapy and Community Reinforcement Approach For Treating Alcohol Problems in the Elderly
Brief Title: Treatment of Alcohol Problems in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kjeld Andersen (Other)
Collaborators: University of New Mexico (Other); Addiction Research Unit, Technische Universität, Dresden, Germany (Other); Institut für Therapieforschung, München, Germany (Unknown)
Responsible Party: Sponsor-Investigator, Kjeld Andersen, Professor, University of Southern Denmark
Organization: University of Southern Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RESCueH-Elderly
Record Dates: First submitted 2014-03-07; First posted 2014-03-11 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Alcohol Use Disorders
Keywords: alcohol; 60+ years; treatment; met; cra; multi site; multi country; questionnaire; random
MeSH Terms: conditions — Alcoholism | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MET (Other): Motivational Enhancement Therapy (MET)
  Interventions: Behavioral: MET + CRA
- MET + CRA (Other): Motivational Enhancement Therapy (MET) with subsequent add-on The Community Reinforcement Approach (CRA)
  Interventions: Behavioral: MET + CRA

INTERVENTIONS:
Behavioral: MET + CRA
  Other Names: Motivational Enhancement Therapy (MET); with subsequent add-on The Community Reinforcement Approach (CRA)

SUMMARY:
With the aging of western societies in the coming years combined with increasing alcohol consumption among elderly, the number of elderly with alcohol problems is expected to rise considerably.

Elderly patients are often lonely; suffer from feelings of loss, fear to be a burden on their children and on society, and feel powerless. On the surface their alcohol related problems seem less severe that those of the middle-aged patients while in reality co-morbidity and social issues complicate alcohol dependency.

Currently, no specific treatment tailored for alcohol use disorder among elderly is available. Consequently they receive either no treatment, are given brief advising from the general practitioner or are referred to treatment at specialized treatment institutions with no specific treatment for elderly.

The investigators propose a study aimed at developing and testing an outpatient behavior therapy program for alcohol use disorders for seniors (60 years and older), which - if effective - can be easily implemented in routine care. Three centers from Denmark, Germany and USA (New Mexico) will participate. All three centers have a long and extensive experience with alcohol treatment and alcohol research. Patients fulfilling the DSM 5 criteria for alcohol use disorder are eligible for the study.

After informed consent participants will be randomly assigned to either Motivational Enhancement Therapy (MET), four sessions/one session per week or MET followed by Community Re-enforcement Approach (CRA), eight sessions/one session per week - thus 12 weeks of treatment in total. 50% will receive MET and 50% MET+CRA. Primary outcome is percentage of patients with abstinence or controlled use (alcohol intake of equivalent blood alcohol content equal to or less than 0.5‰.). A total of 1000 patients will be enrolled. Participants will be assessed with a battery of international validated instruments measuring drinking pattern as well as key elements of treatment.

Participants are assessed before initiation of treatment, at the end of MET treatment (four weeks), at the end of MET+CRA treatment (12 weeks), at 6 months, and at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Seniors (+60 years) with alcohol use disorders according to DSM 5
* Passing an "inclusion quiz" based on 10 questions pertaining to the implications of participating in the study, e.g. knowledge about that it is voluntary to participate, a person declining to participate will receive the standard treatment offered by the treatment clinic, an acceptance of participating can always be withdrawn. The quiz will be conducted after informed consent, and be in a multiple-choice format.

Exclusion Criteria:

* We strive for ecological validity and will only exclude patients who are unable to participate in the therapy or are suffering from severe conditions judged to risking the validity of the study:

  1. 7 or less correct answers in the "inclusion quiz" - indicating cognitive problems or not fully understanding the implications of participating in the study.
  2. Psychotic disorder with positive and/or negative symptoms
  3. Severe depression at time of inclusion
  4. Bipolar disorder
  5. Suicidal thoughts/behaviour at time of inclusion
  6. Use of illicit opioids and/or illicit stimulants (all other forms of medication is allowed, including opioids on prescription - they will be recorded and may be included as covariates in the analyses)
  7. Participating or have participated in other alcohol treatment programs within the last 30 days of inclusion. Pure detoxifications are not an exclusion criteria
  8. Clients with legally authorized representatives

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 704 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Alcohol consumption 26 weeks after baseline | 26 weeks after baseline
  Percentage of patients with abstinence or controlled use (daily alcohol intake equivalent to a BAC equal to or less than 0.5‰) in the last 30 days at 26 weeks after start of treatment. Measured by Form90

SECONDARY OUTCOMES:
Abstinence or controlled use of alcohol | 4 weeks after baseline
  Percentage of patients with abstinence or controlled use (maximum daily alcohol intake of an equivalent of BAC 0.5‰)
  1. In the last 7 days before planned termination of treatment (MET)
Abstinence or controlled use of alcohol | 12 weeks after baseline
  Percentage of patients with abstinence or controlled use (maximum daily alcohol intake of an equivalent of BAC 0.5‰)
  1. In the last 7 days before planned termination of MET + CRA
  2. Participants in MET only, will also be measured
Abstinence or controlled use of alcohol | 52 weeks after baseline
  Percentage of patients with abstinence or controlled use (maximum daily alcohol intake of an equivalent of BAC 0.5‰)
  1. Since 26 weeks follow-up
  2. In the last 30 days at 52 weeks follow-up

OTHER OUTCOMES:
Changes in Quality of life | 52 weeks after baseline
  Quality of life measured by WHO QOL BREF and Personal Happiness Form

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Andersen, MD PhD, Principal Investigator — University of Southern Denmark
Locations (1):
- Unit if Clinical Alcohol Research, Odense, Denmark

REFERENCES:
- [Derived] Behrendt S, Kuerbis A, Braun-Michl B, Bilberg R, Buhringer G, Bogenschutz M, Mejldal A, Andersen K, Sogaard Nielsen A. Residual alcohol use disorder symptoms after treatment predict long-term drinking outcomes in seniors with DSM-5 alcohol use disorder. Alcohol Clin Exp Res. 2021 Nov;45(11):2396-2405. doi: 10.1111/acer.14722. Epub 2021 Oct 9. PMID 34585747
- [Derived] Behrendt S, Kuerbis A, Mejldal A, Braun-Michl B, Bilberg R, Bu Hringer G, Bogenschutz M, Nielsen AS, Andersen K. The Prognostic Role of DSM-5 Alcohol Use Disorder Severity and Age of Onset in Treatment Outcome Among Adults Aged 60. J Addict Med. 2022 May-Jun 01;16(3):303-309. doi: 10.1097/ADM.0000000000000892. PMID 34282079
- [Derived] Mejldal A, Andersen K, Behrendt S, Bilberg R, Christensen AI, Lau CJ, Moller S, Nielsen AS. History of healthcare use and disease burden in older adults with different levels of alcohol use. A register-based cohort study. Alcohol Clin Exp Res. 2021 Jun;45(6):1237-1248. doi: 10.1111/acer.14615. Epub 2021 May 6. PMID 33860951
- [Derived] Mejldal A, Andersen K, Behrendt S, Bilberg R, Bogenschutz M, Braun-Michl B, Buhringer G, Sogaard Nielsen A. Stability of Posttreatment Reductions in World Health Organization (WHO) Drinking Risk Levels and Posttreatment Functioning in Older Adults with DSM-5 Alcohol Use Disorder: Secondary Data Analysis of the Elderly Study. Alcohol Clin Exp Res. 2021 Mar;45(3):638-649. doi: 10.1111/acer.14562. Epub 2021 Mar 3. PMID 33496964
- [Derived] Behrendt S, Kuerbis A, Bilberg R, Braun-Michl B, Mejldal A, Buhringer G, Bogenschutz M, Andersen K, Nielsen AS. Impact of comorbid mental disorders on outcomes of brief outpatient treatment for DSM-5 alcohol use disorder in older adults. J Subst Abuse Treat. 2020 Dec;119:108143. doi: 10.1016/j.jsat.2020.108143. Epub 2020 Oct 5. PMID 33138927
- [Derived] Andersen K, Behrendt S, Bilberg R, Bogenschutz MP, Braun B, Buehringer G, Ekstrom CT, Mejldal A, Petersen AH, Nielsen AS. Evaluation of adding the community reinforcement approach to motivational enhancement therapy for adults aged 60 years and older with DSM-5 alcohol use disorder: a randomized controlled trial. Addiction. 2020 Jan;115(1):69-81. doi: 10.1111/add.14795. Epub 2019 Nov 1. PMID 31454444
- [Derived] Andersen K, Bogenschutz MP, Buhringer G, Behrendt S, Bilberg R, Braun B, Ekstrom CT, Forcehimes A, Lizarraga C, Moyers TB, Nielsen AS. Outpatient treatment of alcohol use disorders among subjects 60+ years: design of a randomized clinical trial conducted in three countries (Elderly Study). BMC Psychiatry. 2015 Nov 14;15:280. doi: 10.1186/s12888-015-0672-x. PMID 26573323